CLINICAL TRIAL: NCT02210273
Title: Evaluation of the Solace Bladder Control System in the Treatment of Female Subjects With Stress Urinary Incontinence
Brief Title: Solace Stress Urinary inContinence Control Efficacy and Safety Study
Acronym: SUCCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solace Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CD1001
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence; SUI
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment (Experimental): Subjects undergoing treatment with the Solace Bladder Control (Vesair) Balloon on day 0
  Interventions: Device: Solace Bladder Control (Vesair) Balloon
- Solace Sham Treatment (Sham Comparator): Subjects undergoing sham treatment on day 0, and treatment with the Solace Bladder Control (Vesair) Balloon at 3 months
  Interventions: Device: Solace Bladder Control (Vesair) Balloon; Device: Solace Sham Treatment

INTERVENTIONS:
Device: Solace Bladder Control (Vesair) Balloon — Subjects may undergo treatment every 12 months until study completion.
  Other Names: Vesair Balloon
Device: Solace Sham Treatment — Sham treatment that resembles treatment with the Solace Bladder Control (Vesair) Balloon
  Arms: Solace Sham Treatment

SUMMARY:
The SUCCESS Trial is designed to determine whether the Solace Bladder Control System is safe and effective for the treatment of Stress Urinary Incontinence (SUI) in adult females.

DETAILED DESCRIPTION:
Subject will undergo treatment with the Solace Bladder Control System or a sham procedure, with the results being compared at 3 months.

All patients undergoing sham treatment are treated at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years of age or older with stress urinary incontinence (SUI)
* Experienced SUI for at least 12 months and attempted and failed prior noninvasive treatment
* Willing to undergo cystoscopic procedures required and 36 month follow-up
* On stable medication for a minimum of 3 months
* Free of local genital skin infection
* Positive Pad Weight Test
* Free of impassable urethral strictures, trauma or necrosis

Exclusion Criteria:

* Pregnant or planning to become pregnant during the study period
* Non-ambulatory or bedridden or physically unable to complete test exercises
* Morbidly obese (defined as BMI ≥ 40 kg/m2)
* Incontinence of neurogenic etiology
* Urge predominant Mixed Incontinence
* Bladder infection (including bladder inflammation or edema) or Urinary Tract Infection (UTI) within 3 months
* History of recurrent urinary tract infections
* Prior surgical procedure for incontinence within the past 6 months
* Is taking medications for urinary incontinence other than anticholinergics
* History of recurrent (>1) or recent (within 5 years) kidney stone(s)
* Has a prosthetic heart valve
* Unable to tolerate any form of antibiotic
* Taking anticoagulation therapy, other than aspirin
* Has urinary incontinence due to Intrinsic Sphincter Deficiency (ISD)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-08-11 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Improvement in quality of life as assessed by pad weight tests assessments and questionnaires | 3 Months
  Comparison of increases in pad weight test and patient reported outcomes on questionnaires

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events | 3 Months
  Site-reported adverse events designated as related to the treatment
Severity of treatment-related adverse events | 3 Months
  Site-reported adverse events designated as related to the treatment.

OTHER OUTCOMES:
Improvement in quality of life in all patients assessed with pad weight tests and questionnaires | 36 Months
  Comparison of increases in pad weight test and patient reported outcomes on questionnaires
Severity of all adverse events | 36 Months
  Site-reported adverse events designated as related to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rovner, MD, Principal Investigator — Medical University of South Carolina
Locations (20):
- United States (20):
  - Valley Urogynecology Associates, Phoenix, Arizona
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Urology Associates of Norwalk, Norwalk, Connecticut
  - WomanCare, Arlington Heights, Illinois
  - Women's Health Institute of Illinois, Oak Lawn, Illinois
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology, Glen Burnie, Maryland
  - Chesapeake Urology, Owings Mills, Maryland
  - Female Pelvic Medicine and Urogynecology Institute of Michigan, Grand Rapids, Michigan
  - North Shore LIJ, Great Neck, New York
  - Premier Medical Group, Newburgh, New York
  - Premier Medical Group, Poughkeepsie, New York
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Women and Infants Hospital, Providence, Rhode Island
  - MUSC Urology, Charleston, South Carolina
  - Sanford Female Pelvic Medicine and Reconstructive Surgery Clinic, Sioux Falls, South Dakota
  - Virginia Women's Center, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - Integrity Medical Research, Mountlake Terrace, Washington

IPD SHARING:
Plan to Share IPD: No
Individual records will not be made available to honor contracts with Investigators.

REFERENCES:
- [Derived] McCammon K, Jacoby K, Kalota S, Snyder J, Cline K, Robertson K, Rardin C, Kahan R, Green L, Zuckerman J, Rovner E. Three-month primary efficacy data for the SUCCESS Trial; a phase III, multi-center, prospective, randomized, controlled study treating female stress urinary incontinence with the vesair intravesical balloon. Neurourol Urodyn. 2018 Jan;37(1):440-448. doi: 10.1002/nau.23324. Epub 2017 Nov 2. PMID 29095516